CLINICAL TRIAL: NCT04100980
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Chronic Urinary Tract Infections (UTI)
Status: Withdrawn | Type: Observational
Why Stopped: Company shifted focus
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-014
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic UTI; Chronic Urinary Tract Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic UTI: Patients who have been diagnosed with chronic urinary tract infections (UTI).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study

SUMMARY:
Correlation of Microbiome to Chronic Urinary Tract Infections (UTI) via Relative Abundance Found in Microbiome Sequencing

DETAILED DESCRIPTION:
Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific Chronic UTI types.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient
2. Male or female patients age 18 and older.
3. Diagnosis of chronic UTIs by a physician based upon urinalysis and/or urine culture.

Exclusion Criteria:

1. Refusal by patient to sign informed consent form
2. Treatment with antibiotics within 2 weeks prior to screening
3. Treatment with probiotics within 6 weeks prior to screening
4. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
5. Postoperative stoma, ostomy, or ileoanal pouch
6. Participation in any experimental drug protocol within the past 12 weeks
7. Treatment with total parenteral nutrition
8. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
9. Inability of patient to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have been diagnosed with chronic urinary tract infections (UTI)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to chronic Urinary Tract Infection (UTI) via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific chronic urinary tract infection (UTI) types.

SECONDARY OUTCOMES:
Validation of Sequencing Methods | 1 year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only aggregated and deidentified data will be shared with other researchers.